CLINICAL TRIAL: NCT01169311
Title: A Prospective, Multi-Center Investigation Of The Safety And Performance Of The Covidien EEA™ Hemorrhoid And Prolapse Stapling Set With DST Series™ Technology Im A Hemorrhoidopexy Procedure
Brief Title: Safety and Performance of the Covidien EEA Hemorrhoid and Prolapse Stapling Set in a Hemorrhoidopexy Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVHEPH0021
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Hemorrhoid
Keywords: Hemorrhoids; Hemorrhoid; grade II, III, IV
MeSH Terms: conditions — Hemorrhoids; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HEEA Stapler (Experimental): hemorrhoidopexy using Covidien EEA Hemorrhoid and Prolapse Stapling Set
  Interventions: Device: Hemorrhoidopexy

INTERVENTIONS:
Device: Hemorrhoidopexy
  Other Names: Covidien EEA Hemorrhoid and Prolapse Stapling set

SUMMARY:
Trial Objectives

The primary objectives of this clinical trial are to estimate the Covidien EEA™ Hemorrhoid and Prolapse Stapling Set:

overall performance defined by the successful creation of a normal staple line safety as measured by the 30 day incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign Informed Consent Form
* The participant must be 18-80 years of age.
* The participant has (symptomatic) Grade 2-4 Hemorrhoids and is eligible for stapled hemorrhoidopexy.

Exclusion Criteria:

* The procedure is needed as revision hemorrhoid surgery.
* The participant is pregnant.
* The participant has an active or a history of infection requiring antibiotics at the intended operative site within thirty (30) days prior to the planned surgery date.
* The participant is unable or unwilling to comply with the study requirements, follow-up schedule.
* The participant has a history of drug or alcohol abuse.
* The participant has a history of venous thrombosis or pulmonary embolism.
* The participant has a history of coagulopathy.
* The participant is taking aspirin, anti-coagulation and/or anti platelet therapies (e.g.: Warfarin, Levonox) within the last 7 days prior to the planned surgery date
* The participant has a history of fecal incontinence.
* The participant has co-morbidities which, in the opinion of the investigator, will not be appropriate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Lee, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 21 July 2010 and 17 March 2011 patients were recruited at 2 medical clinic and one hospital; subjects with grades 2-4 hemorrhoids eligible for stapled hemorroidopexy were assessed for eligibility for study; exclusion criteria: pregnant,Ab use for SSI, drug/alcohol abuse, aspirin/anticuagulant therapy, hx VT, hx PE,
Groups:
- Covidien EEA Hemorrhoid and Prolapse Stapler: Subjects meeting inclusion/exclusion criteria will undergo hemorrhoidopexy with the Covidien EEA hemorrhoid and prolapse stapler set.
Period: Overall Study
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Covidien EEA Hemorrhoid and Prolapse Stapler: Subjects undergoing hemorrhoidopexy with HEEA stapler
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Uneventful Creation of a Functional Staple Line at First Firing of Device
Description: Successful creation of staple line at first firing of device during hemorrhoidopexy
Time Frame: about 20 minutes for procedure
Measure: Number; unit: participants
Groups:
- Covidien EEA Hemorrhoid and Prolapse Stapler: subjects will have have hemorrhoidopexy using the EEA stapler
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 27
participants | 27

2. Secondary Outcome: OR Time
Description: Duration of procedure
Time Frame: Day 0 - Time of stop minus time of start
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 27
minutes | 21.5 (7.8)

3. Secondary Outcome: Intra-Operative Bleeding Requiring Intervention
Description: Incidence of intervention for intra-operative staple-line bleeding
Time Frame: Day 0 - time of surgery
Measure: Number; unit: participants
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 27
participants | 12

4. Secondary Outcome: Length of Stay
Description: length of time between time of admission and time of discharge
Time Frame: Day 0, time of discharge minus time of admission
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 27
Minutes | 146.6 (167.5)

5. Secondary Outcome: Time to Return to Normal Activity
Time Frame: 30 days post op
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 27
Days | 11.1 (5.5)

6. Secondary Outcome: Incidence of Stapler Malfunction or Misfires
Time Frame: about 20 minutes for procedure
Measure: Number; unit: participants
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 27
participants | 0

7. Secondary Outcome: Post Operative Pain
Description: Post operative pain measured by 11 point visual analog scale, measured as change from baseline The scale range is 0-10, where 0 = no pain and 10 = worst possible pain
Time Frame: baseline, 30 days post op
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 27
units on a scale | -1.0 (1.5)

8. Secondary Outcome: Quality of Life, Physical Component
Description: Physical component score SF36 scale measured as change from baseline the scoring ranges from 0 to 100 with 0 = unable to do anything while 100 = capable of physical activity without limitation
Time Frame: baseline, 30 days post op
Population: Only subjects who completed the SF-36 questionnaire were included in the analysis. The number of participants reflects 24/27 subjects completed the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 24
units on a scale
  Baseline | 52.95 (8.00)
  30 days post op | -1.61 (8.33)

9. Secondary Outcome: Quality of Life, Mental Component
Description: quality of life, SF36 measure as change from baseline the scoring ranges from 0 to 100 with 0 = complete mental activity limitation; while 100 = capable of mental activity without limitation
Time Frame: Baseline, 30 days post op
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Number analyzed (Participants) | 24
units on a scale
  Baseline | 56.12 (5.47)
  30 Days post op | -0.07 (3.74)

ADVERSE EVENTS:
Time Frame: Adverse events were colllected from time of enrollment (Day 0, time of surgery) until subject's final visit at one month +/- 1 week post surgery.
Arm/Group | Covidien EEA Hemorrhoid and Prolapse Stapler
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 15/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Covidien EEA Hemorrhoid and Prolapse Stapler (N=27)
Anorectal Discomfort (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
proctalgia (Gastrointestinal disorders) | 9
Rectal Hemorrhage (Gastrointestinal disorders) | 11
vomitting (Gastrointestinal disorders) | 2
Local Swelling (General disorders) | 2
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No